CLINICAL TRIAL: NCT00553124
Title: Bladder Cancer Prognosis Programme (Incorporating SELENIB Trial)
Brief Title: Different Factors Affecting Patients With Newly Diagnosed Bladder Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Prevention
Other Study IDs: CDR0000572089; CRUK-BCPP-2005-01; ISRCTN13889738; EU-20768
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2007-10

CONDITIONS: Bladder Cancer
Keywords: stage 0 bladder cancer; stage I bladder cancer; stage II bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Selenium; Vitamin E; Biopsy; Chemoprevention; Cryopreservation; Gene Expression Profiling; Immunohistochemistry; Polymerase Chain Reaction

INTERVENTIONS:
Drug: selenium
Drug: vitamin E
Procedure: biopsy
Procedure: chemoprevention
Procedure: cryopreservation
Procedure: cytology specimen collection procedure
Procedure: diagnostic procedure
Procedure: gene expression analysis
Procedure: immunohistochemistry staining method
Procedure: laboratory biomarker analysis
Procedure: medical chart review
Procedure: mutation analysis
Procedure: polymerase chain reaction
Procedure: quality-of-life assessment
Procedure: questionnaire administration
Procedure: study of socioeconomic and demographic variables

SUMMARY:
RATIONALE: Studying different factors that effect patients with newly diagnosed bladder cancer may help doctors learn more about the disease, improve the ability to plan cancer treatment, and help patients live more comfortably.

PURPOSE: This clinical trial is studying different factors affecting patients with newly diagnosed bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the effect of lifestyle factors (e.g., smoking, dietary habits, fluid intake, or environmental exposures) on the recurrence and progression of bladder cancer.
* To assess the impact of selenium and/or vitamin E on the progression and recurrence of bladder cancer.
* To study health-related quality of life and its association with recurrence and progression of bladder cancer.
* To establish a bladder cancer tissue bank that will comprise blood, urine, and bladder tissue.
* To study the predictive effect of molecular markers on the recurrence and progression of bladder cancer.

OUTLINE: This is a multicenter study.

The study will be based on a cohort of patients with newly detected bladder cancer in all 16 urological centres within the West Midlands, commencing in late 2005 for a period of 5 years. This research project consists of 5 individual studies: CRUK-BCPP-2005-01-COHORT, CRUK-BCPP-2005-01-MARKERS, CRUK-BCPP-2005-01-QOL, CRUK-BCPP-2005-01-TISSUE-BANK, and CRUK-BCPP-2005-01-TREATMENT. Patients may participate in all or only some of these individual studies.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Bladder lesion with cystoscopic characteristics compatible with urothelial cancer or transitional cell carcinoma meeting 1 of the following criteria:

  * Non-muscle-invasive tumor
  * Muscle-invasive tumor
  * Solitary G1 pTa tumor
* No previous diagnosis of cancer of the urethra, bladder, ureter, or renal pelvis within the 10 years prior to current diagnosis

PATIENT CHARACTERISTICS:

* Fit for cystoscopy and surgical biopsy/resection
* No HIV infection
* No condition that, in the opinion of the local investigator, might interfere with the safety of the patient or evaluation of the study objectives

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3400
Dates: Start 2005-12

PRIMARY OUTCOMES:
Recurrence-free interval
Progression-free interval

SECONDARY OUTCOMES:
Overall survival time
Incidence of transitional cell carcinoma outside the bladder
Incidence of all other malignancies clinically diagnosed
Incidence of cardiovascular events
Quality of life as measured by EORTC QLQ-C30, QLQ-BLS24 and QLQ-BLM30 questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: K. K. Cheng, MD, Study Chair — University Hospital Birmingham
Locations (1):
- Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England, United Kingdom